CLINICAL TRIAL: NCT04359225
Title: A Comparison of 3D and 2D Telemedicine: Communication During Covid 19
Brief Title: A Comparison of 3D and 2D Telemedicine During Covid 19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Strathclyde (Other); Glasgow Royal Infirmary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: GN20HS182
Record Dates: First submitted 2020-04-16; First posted 2020-04-24 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Telehealth
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patient will be blinded to form of telemedicine. Clinician will not be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D telemedicine (Active Comparator): 3D telemedicine system
  Interventions: Other: 3D Telemedicine
- 2D telemedicine (Placebo Comparator): 2D telemedicine system (standard care)
  Interventions: Other: 2D Telemedicine

INTERVENTIONS:
Other: 3D Telemedicine — Telemedicine using 3D broadcast to clinician
  Other Names: Telepresence
  Arms: 3D telemedicine
Other: 2D Telemedicine — Standard care with 2D telemedicine
  Other Names: Standard Care
  Arms: 2D telemedicine

SUMMARY:
It is critical to establish an effective form of telemedicine during the Covid 19 pandemic, that will allow safe social distancing of clinicians and patients. The investigators serve as the regional plastic, burns and reconstructive centre for the West of Scotland, population 3 million. All face to face clinics have been cancelled and converted to telephone/telemedicine only consultations. The investigators will establish both 2D and 3D telemedicine as normal patient follow up practice during this period.

The aim is to implement a 3D telemedicine system to facilitate patient follow up and remote physiotherapy, that will act as if the patient is physically 'present' in the room. Physiotherapy is crucial to patient outcomes after burns contractures, hand trauma and cancer reconstruction. The 3D telemedicine system will be built by an industrial partner, with CE marked equipment, specifically to help during the Covid-19 Pandemic.

This study forms a follow on study to the investigator's pilot study (based on clinical feedback only)

DETAILED DESCRIPTION:
During Covid pandemic the Canniesburn Plastic Surgery Unit has stopped face to face clinics. The investigators therefore aim to assess current telemedicine options from a clinician viewpoint.

Why is the 3D telemedicine study important during Covid 19?

1. Augment not replace current telemedicine capabilities. 3D telemedicine system would be transformative - much of Plastic Surgery work is 3 dimensional e.g. burns contractures, cleft lip. A 3D system may therefore give clinicians a more 'realistic' and accurate representation of patient interaction.
2. Reduce viral load in clinic. This will reduce face to face contact. High viral load transmission (eg in the confines of an all day clinic) may be associated with higher risk of healthcare worker mortality.
3. Facilitate remote therapies and improve patient outcomes. Current 2D telemedicine (e.g. Attend Anywhere) is limited in the ability to remotely guide patient therapies - the therapist cannot guide the camera or look at specific areas of interest. With 3D telemedicine the therapist can 'walk around' the patient as if the patient were co-present, and look at areas of interest with ease.
4. Measurements of angles/other clinical measurements. For example, after a burns contracture or hand trauma a clinician may want to measure the angles at the wrist joint to see if there is any improvement. This cannot be done accurately with 2D telemedicine. 3D telemedicine may facilitate the measurement of angles and assess outcomes but this is unknown.

Method Randomised Controlled Trial. Single blinded (participants blinded - unaware of type of telemedicine, clinicians unblinded - aware of type of telemedicine)

Study setting and Participants:

The study will review clinician's assessments of telemedicine and clinical assessment of patients using telemedicine. These will consist of the plastic surgery patients selected from general plastic surgery clinic including patients with breast reconstruction, sarcoma, limb reconstruction, head & neck reconstruction, flap reconstruction, hand trauma and cleft lip, and will be known to the research team. The assessment is of the telemedicine system by the clinician only. There will be two sites, the 'remote' site where the patient attends, and the 'central' site where the clinician reviews the patient. Remote site will be at West Glasgow Ambulatory Care Hospital (Covid free site) and the central location will be Glasgow Royal Infirmary.

Outcomes The investigators aim to answer the question "How does 3D telemedicine compare to 2D telemedicine?"

Primary outcomes:

Mental Effort Rating Scale, University Hospital of North Norway (UNN) scales, Telehealth Usability Questionnaire (TUQ)

Secondary outcomes:

Subjective feedback with transcribing, coding and thematic analysis. Measurements (where applicable e.g. angles of contracture in hand) Outcome scoring scales (where applicable e.g. validated Unilateral Cleft Score Surgical Outcomes Evaluation Scale - UCLSOE).

Study Methods:

Sample Size The pilot/feasibility study will generate data for sample size calculation. No data exist for sample size calculations of 3D versus 2D telemedicine.

Randomisation Block randomisation. Patient randomised to 2D or 3D telemedicine first.

Patient assessment with Telemedicine The patient is examined with the randomly allocated type of telemedicine and the duration of consultation recorded. The telemedicine room is the same for both 2D and 3D telemedicine, and uses the same equipment. After the consultation the patient does not require further participation

Clinician Feedback The clinician fills in a questionnaire assessment of the type of telemedicine used.

Clinician records measurements where applicable Clinician records outcome scoring scales where applicable

Primary outcomes UNN questionnaire Mental Effort Rating Scale

Secondary outcomes Telehealth Usability Questionnaire Subjective interview Patient measurements (where applicable) Patient outcome scales (where applicable)

ELIGIBILITY:
Inclusion Criteria:

* Breast reconstruction patients pre and post op
* Sarcoma patients pre and post op
* Burns patients pre and post op
* Cleft lip patients pre and post op
* Head & neck reconstruction patients pre and post op
* Hand trauma patients pre and post op
* Flap reconstruction patients pre and post op.

Exclusion Criteria:

* Adults unable to consent
* Patients requiring interpreter.

Ages: 1 Year to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-30 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
University Hospitals of North Northway questionnaire | Single time point at day 1 (Clinician assesses telemedicine system once after seeing patient)
  University Hospitals of North Northway questionnaire. Outcome scale with a sum score 1 to 5 Higher score is worse
Mental effort rating scale | Single time point at day 1(Clinician assesses telemedicine system once after seeing patient)
  Scale 1 to 9 Higher score is worse

SECONDARY OUTCOMES:
Telehealth Usability Questionnaire | Single time point at day 1 (Clinician assesses telemedicine system once after seeing patient)
  Telehealth Usability Questionnaire. 21 domains, each with scale 1 to 7. Higher is better.
Subjective feedback interview | Once at study completion, an average of 18 months.
  Clinician Subjective feedback. This is an interview performed by a psychologist and will be transcribed, coded and thematically analysed. There is no statistical analysis or outcome scale involved.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lo, FRCS Plast, Principal Investigator — NHS Greater Glasgow and Clyde Clinical Research and Development Central Office
Locations (1):
- Canniesburn Regional Plastic Surgery and Burns Unit, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No